CLINICAL TRIAL: NCT04945161
Title: A Randomized, Double-blind, Placebo-controlled Clinical Study to Explore the Mechanism of Action (MOA) of ON101 Cream in Patients With Diabetic Foot Ulcers (DFUs).
Brief Title: A Randomized,Double-blind,Placebo-controlled Clinical Study to Explore the Mechanism of Action of ON101 Cream in Patients With DFUs.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ON101CLIIS01-DFU
Record Dates: First submitted 2021-03-22; First posted 2021-06-30 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled clinical study to explore the mechanism of action (MOA) of ON101 cream in patients with diabetic foot ulcers (DFUs).The primary objective is to explore the mechanistic role of ON101 cream in healing diabetic foot ulcers by determining the molecular targets of ON101 cream.
Who Masked: Participant, Investigator
Masking Description: Study design:
  1. □Control: ■placebo
     * active (please specify name and dosage)
     * other
     * Uncontrolled
  2. Blinding: □open-label □evaluator blind □single blind ■double blind
     □double dummy □other
  3. Randomized: ■yes □no
  4. ■Parallel □Cross-over □Other
  5. Duration of treatment: Six (6) weeks
  6. Titration: □forced □optional ■none
  7. □Multi-national ■Multi-center(Taiwan): 2 sites □Single center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: N = 6 ON101 plus SoC (Experimental): Twelve (12) eligible subjects with DFUs will be enrolled. These 12 subjects will be randomly assigned to receive either ON101 treatment plus SoC (Arm A) or Placebo plus SoC (Arm B) for six weeks. Treatment arm allocation will be done through randomization in a double-blind fashion.
  SoC will be provided from screening to the end of treatment. The SoC includes evaluation to ensure adequate arterial flow, wound cleaning, removal of necrotic, infected and/or nonviable tissue by debridement, maintenance of moist wound environment via regular changing of dressings, and management of infection through oral antibiotics, if necessary.
  Interventions: Drug: ON101 Cream
- Arm B: N = 6 Placebo plus SoC (Placebo Comparator): Twelve (12) eligible subjects with DFUs will be enrolled. These 12 subjects will be randomly assigned to receive either ON101 treatment plus SoC (Arm A) or Placebo plus SoC (Arm B) for six weeks. Treatment arm allocation will be done through randomization in a double-blind fashion.
  SoC will be provided from screening to the end of treatment. The SoC includes evaluation to ensure adequate arterial flow, wound cleaning, removal of necrotic, infected and/or nonviable tissue by debridement, maintenance of moist wound environment via regular changing of dressings, and management of infection through oral antibiotics, if necessary.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ON101 Cream — Active ingredients: Extracts of Plectranthus amboinicus and Centella Asiatica
  Arms: Arm A: N = 6 ON101 plus SoC
Other: Placebo — Placebo
  Arms: Arm B: N = 6 Placebo plus SoC

SUMMARY:
The primary objective is to explore the mechanistic role of ON101 cream in healing diabetic foot ulcers by determining the molecular targets of ON101 cream.

Primary endpoint:

Percentage change from baseline in the expression level of individual target gene(s) at protein and/or mRNA level.

Secondary endpoints:

1. Comparison of the gene and/or protein expression level of individual target between ON101 and Placebo groups
2. Change from baseline in the wound microbiota composition in each group
3. Comparison of the wound microbiota composition between ON101 and Placebo groups
4. Comparison of the wound reduction rate in each group
5. Correlation of wound reduction rate with the alternated level of each target gene in each group.

Safety endpoints:

Incidence of treatment-emergent adverse event (AE) Change from baseline in vital signs, physical examination, and laboratory tests

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study to explore the mechanism of action (MOA) of ON101 in treating chronic diabetic foot ulcers (DFUs). There will be 6 subjects ON101 treatment (Arm A) and 6 subjects in Placebo (Arm B) .

Twelve(12) eligible subjects with DFUs and are not undergoing dialysis will be enrolled and randomly assigned to receive either ON101 treatment (Arm A) or Placebo (Arm B) for six weeks. Treatment arm allocation will be done through randomization in a double-blind fashion. SoC will be provided throughout the study period.Subjects with DFUs not undergoing dialysis, N = 12 Arm A: ON101 plus SoC, N = 6 Arm B: Placebo plus SoC, N =6 SoC will be provided throughout the study period (from screening to end of treatment). SoC includes evaluation to ensure adequate arterial flow, wound cleaning, removal of necrotic, infected and/or nonviable tissue by debridement, maintenance of moist wound environment via regular changing of dressings, and management of infection through oral antibiotics, if necessary.

The study will have three periods, a Screening/Run-in Period, a Treatment Period, and a Safety Follow-up Period.

Screening/Run-in Period (14 days):

Treatment Period (up to 6 weeks ± allow window):

There will be five (5) visits during the Treatment Period. Baseline/V1 (Day 1 ± 3 days) Visit 2 to Visit 5/EOT (Day 14 to Day 42/EOT) Safety Follow-up Period (Day 49±1 or Day of EOT + 6-8 days)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, male or female, aged 20 to 80 years (inclusive) with Type 1 or Type 2 diabetes undergoing therapy for glycemic control.
2. Subjects has a glycosylated hemoglobin, HbA1c < 12%.
3. Presence of at least one diabetic foot ulcer that meets all of the following criteria:

   1. At the time of Visit 0 (V0), the ulcer has existed for at least one month;
   2. At the time of Visit 1 (V1), the post-debridement ulcer presents Grade 2 or Grade 3 (without osteomyelitis or active infection) in Wagner Ulcer Classification System assessment; and
   3. Area should be ≥ 4 cm2 and ≤ 25 cm2;
   4. No higher than the ankle.
4. Subject has adequate vascular perfusion of the affected limb, confirmed by Ankle-Brachial Index (ABI) ≥ 0.8 and ≤ 1.3.
5. Clinically normal resting ECG at the first Screening Visit (V0) or, if abnormal, considered to be not clinically significant by the Investigator.
6. Subject must use an off-loading method for the target ulcer on the plantar during the whole study period.
7. Subject, if female of child-bearing potential, has a negative pregnancy test on urine at screening, must not be breastfeeding, and willing to use two medically accepted methods of contraception (e.g., barrier contraceptives [female condom or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptives rings], and intrauterine devices) during the course of the study (excluding women who are not of childbearing potential and/or who have been sterilized).
8. Subject is able and willing to comply with the study procedures.
9. A signed and dated informed consent form has been obtained from the subject.

Exclusion Criteria:

1. In response to standard of care (SoC), ulcer size reduction is ≥20% during the two-week run-in screening period (between the first Screening Visit/V0 and Baseline Visit/V1).
2. Ulcers with exposed bone or associated with osteomyelitis. Note: The osteomyelitis should be ruled out by clinical examination (probing of the wound) or X-ray findings where find necessary by the Investigator.
3. Presence of necrosis, purulence, or sinus tracts that cannot be removed by debridement.
4. Laboratory values at Screening of:

   1. Liver function test (total bilirubin, aspartate aminotransferase [AST], or alanine transaminase [ALT]) > 3x the upper limit of normal, or
   2. Albumin < 2.5 g/dL, or
   3. Renal function test (serum creatinine or urea) > 2x the upper limit of normal
5. Presence of any clinically significant medical condition(s) in medical history during screening period that, in the opinion of the Investigator, could interfere with wound healing, including but not limited to the following:

   1. Acute or unstable Charcot foot
   2. Current sepsis
   3. Active malignant disease. A subject, who has had a malignant disease in the past, was treated and is currently disease-free, maybe considered for study entry.
   4. Acquired immune deficiency syndrome (AIDS) or HIV positive
6. Subject is currently receiving (i.e., within 30 days of randomization visit) or scheduled to receive any of the following medication or therapies, could interfere with wound healing during the course of the study:

   1. Immunosuppressive or chemotherapeutic agents, radiotherapy, or systemic corticosteroids
   2. Autoimmune disease therapy
   3. Lower limb revascularization surgery (e.g., angioplasty, artery bypass surgery)
   4. Hyperbaric oxygen therapy
   5. Bioengineered tissue or skin substitutes
   6. Use of any investigational drug(s)
   7. Cell therapy
7. More than two (2) ulcers located on or below the malleoli on the target foot.
8. A psychiatric condition (e.g., suicidal ideation), current or chronic alcohol or drug abuse problem, determined from the subject's medical history, which in the opinion of the Investigator, may pose a threat to subject compliance.
9. Has any other factor which may, in the opinion of the Investigator, compromise participation and/or follow-up in the study.
10. Body mass index (BMI) >40 with plantar ulcer.
11. Heavy smoker (>1 pack per day).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Primary endpoint:Q-RT-PCR, for the inflammation stage and the remodeling stage | Through study completion, an average of 1 year
  Percentage change from baseline in the expression level of individual target gene(s) at protein and/or mRNA level, usch as Q-RT-PCR, Cytokine, Chmokine, GFs.

SECONDARY OUTCOMES:
Secondary endpoint (1): IL-1b, IL-6, TNF, TGF, CXCL9, FGF2, and IL1RN!..ect. | Based on each visit window for the first review, and through study completion, an average of 1 year for the final review
  Comparison of the gene and/or protein expression level of individual target between ON101 and Placebo groups, through Q-RT-PCR, between inflammation stage and remodeling stage
Secondary endpoint (2): iNOS, CD86, CD80, CD163, CD206, KRT14, MMP12..ect. | Based on each visit window for the first review, and through study completion, an average of 1 year for the final review
  Change from baseline in the wound microbiota composition in each group, through IHC, analysis macrophage marker, epithelization, fibroblast maker, collagen, EPC and angiogenesis
Secondary endpoint (3): CO15A1, CD71, CD34..ect | Based on each visit window for the first review, and through study completion, an average of 1 year for the final review
  Comparison of the wound microbiota composition between ON101 and Placebo groups, through IHC, between inflammation stage and remodeling stage.
Secondary endpoint (4):target ulcer size evaluation report (Area: perimeter, length, width ) | Based on each visit window for the first review, and through study completion, an average of 1 year for the final review
  Comparison of the wound reduction rate in each group,through target ulcer size evaluation report (Area: perimeter, length, width )
Secondary endpoint (5): wound reduction rate of each target gene in each group | Based on each visit window for the first review, and through study completion, an average of 1 year for the final review
  Correlation of wound reduction rate with the alternated level of each target gene in each group, through IHC and target ulcer report.

OTHER OUTCOMES:
Safety endpoint(1): Change from baseline in vital signs | Based on each visit window for the first review, and through study completion, an average of 1 year for the final review
  Incidence of treatment-emergent adverse event (AE) Change from baseline in vital signs:pulse rate(times/min), SBP/DBP(mmHg), Body Temperature ( C), and respiratory rate ( breaths/min)
Safety endpoint(2): Change from baseline in physical examination | Based on each visit window for the first review, and through study completion, an average of 1 year for the final review
  Incidence of treatment-emergent adverse event (AE) Change from baseline in physical examination: Heent ( head, eye,ear, nose, throat), Month, Skin, Neck ( including thyroid), Lymph nodes, spine,Cardiovascular system, GI, Nervous, Musculoskeletal, blood, and mental status.
Safety endpoint(3):Change from baseline in laboratory tests | Based on each visit window for the first review, and through study completion, an average of 1 year for the final review
  Incidence of treatment-emergent adverse event (AE) Change from baseline in laboratory tests: Complete blood count (WBC, Neutrophils, Monocytes, Hb, MCV,MCH,MCHC, Platelet), and Biochemistry ( HbA1c, HDL-C, LDL-C, ALT, AST, Creatinine, Albumin, Urea)

CONTACTS AND LOCATIONS:
Locations (1):
- Kueiho Chen, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
IIS study